CLINICAL TRIAL: NCT06730113
Title: Youth-onset Type 2 Diabetes and Heart Disease: The Young at Heart Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001819; 001819-DK
Record Dates: First submitted 2024-12-11; First posted 2024-12-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01-23

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Cardiovascular Disease; Overweight; Obesity; Youth Onset Type 2 Diabetes; Lean
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control lean participants (Y-Lean): A prospective, observational study design in youth aged 12-25 years to compare Y-T2DM with age and BMI-matched youth with overweight or obesity (Y-OW) and age-matched healthy lean peers (Y-Lean).
- Y-T2DM: A prospective, observational study design in youth aged 12-25 years to compare Y-T2DM with age and BMI-matched youth with overweight or obesity (Y-OW) and age-matched healthy lean peers (Y-Lean).
- Youth with overweight/ obesity (Y-OW: A prospective, observational study design in youth aged 12-25 years to compare Y-T2DM with age and BMI-matched youth with overweight or obesity (Y-OW) and age-matched healthy lean peers (Y-Lean).

SUMMARY:
Background:

Type 2 diabetes is a disease that affects blood sugar levels. Complications can include heart and blood vessel (vascular) diseases. Rates of type 2 diabetes have tripled in children and young adults over the last 40 years. Vascular diseases are also increasing in young people.

Objective:

To learn more about factors, including type 2 diabetes, that may cause vascular disease in young people.

Eligibility:

People aged 12 to 25 years who (1) have type 2 diabetes; (2) are overweight but not diabetic; (3) or are lean and healthy. Biological parents are also needed.

Design:

Young participants will visit the NIH clinic once a year for up to 25 years. Each visit will take 4 days. Before each visit, participants will wear devices to track their sleep, activity, and blood sugar levels for 7 to 10 days.

At each visit, participants will have tests including:

Samples: They will provide blood, urine, and stool samples.

Heart: They will ride a stationary bike for 6 minutes with stickers applied to their chest.

Scans: They will lie on a bed that slides into a tube; the machine will take pictures of the inside of their body.

Energy: They will wear a hood over their head to measure the air they breathe.

Social stress: They will give a speech for 10 minutes to show their body s response to stress.

Glucose: They will drink a sweet drink to see how their blood sugar changes.

Biological parents will have 1 study visit. They will have blood tests. They will fill in questionnaires about their lifestyle and stress.

...

DETAILED DESCRIPTION:
Study Description:

This study will evaluate the pathophysiological features of cardiovascular disease in youth-onset type 2 diabetes (Y-T2DM) using a multi-level, multi-domain approach of socio-ecological risk factors (societal, community, and individual). We will employ a prospective, observational study design in youth aged 12-25 years to compare Y-T2DM with age and BMI-matched youth with overweight or obesity (Y-OW) and age-matched healthy lean peers (Y-Lean). The study will also include a single-day visit for biological parents of enrolled Y-T2DM, Y-OW and Y- lean, to assess parental factors involved in the pathophysiology of cardiovascular disease in Y-T2DM.

Objectives:

Primary Objectives:

* To compare pulse wave velocity (PWV) at baseline in Y-T2DM vs Y-OW and age-matched peers Y-Lean.
* To compare augmentation index (Aix) at baseline in Y-T2DM vs Y-OW and age-matched peers Y-Lean.
* To compare pulse wave velocity (PWV) at 5 years in Y-T2DM vs Y-OW and age-matched peers Y-Lean.
* To compare augmentation index (Aix) at 5 years in Y-T2DM vs Y-OW and age-matched peers Y-Lean.

Secondary Objectives:

In Y-T2DM vs. Y-OW vs. Y-Lean youth,

* To evaluate coronary artery structure and endothelial function at baseline and 5 years.
* To evaluate the relationship of pulse wave velocity and coronary artery structure & endothelial function with atherogenic and remnant lipoproteins.

Exploratory Objectives:

In Y-T2DM vs. Y-OW vs. Y-Lean youth,

* To evaluate annual change in vascular aging (measured by the change in pulse wave velocity and endothelial function).
* To evaluate the relationship of physiologic, psychological stress (measured with the allostatic load score, ALS), psychosocial and behavioral factors with vascular aging.
* To evaluate biomarkers for vascular aging; ex. Beta-cell function, insulin resistance, inflammatory markers, and novel lipid parameters.
* To evaluate the association of polygenic risk scores (PRS) in Y-T2DM and with changes in glucose and metabolic profiles (e.g., triglycerides) over time.
* To evaluate differences in epigenetic aging in youth and parents.
* To determine the prevalence rates of major adverse cardiovascular events (MACE)

Endpoints:

Primary Endpoint:

* Carotid-femoral pulse wave velocity (PWV) at baseline
* Pulse augmentation index (Aix) at baseline
* Carotid-femoral PWV at 5 years
* Pulse Aix at 5 years

Secondary Endpoints:

* Right coronary wall thickness measured by cardiac MRI
* Endothelial function measured by MRI isometric handgrip exercise
* Fasting and postprandial lipoprotein profile (mixed meal test)

Exploratory Endpoints:

Markers of vascular aging (annual change):

* PWV
* Aix
* Endothelial function measured by reactive hyperemia index
* Right coronary wall thickness measured by MRI
* Heart rate variability
* Central Retinal Artery Equivalent

Markers of physiological stress

* Allostatic load score
* Cortisol (serum)
* C-reactive protein and immune biomarkers

Assessment of metabolic variables

* Sigma and insulin sensitivity index (standard 75g OGTT)
* Postprandial lipoproteins (mixed meal test)
* Metabolomics, Lipidomics, Proteomics Measures
* Liver fat and function
* Body composition

Psychosocial, Neighborhood, and individual variables

* Psychosocial Assessments: Binge Eating Disorder Screener-7 (BED-7), Brief Resilience Scale, Diabetes Distress Scale (DDS-17), Emotional Eating Scale, Michigan Neuropathy Screening Instrument (MNSI), PROMIS Emotional Distress - Anxiety, PROMIS Emotional Distress - Depression, PROMIS - Sleep Disturbance, Reward-Based Eating Drive Scale (REDS), Self-assessment of Worries, Concerns, and Burdens Related to Diabetes and Preparation for Transitioning, Substance Use, and Stroop Color and Word Test
* Neighborhood Assessments: Adverse Childhood Experience (ACE), Confusion, Hubbub, and Order Scale (CHAOS), MacArthur Scale of Subjective Social Status, Neighborhood Disadvantage Scale, Pediatric ACES and Related Life Events Screening (PEARLS), Unpredictability Beliefs Scale, and U.S. Household Food Insecurity Module.
* Individual Assessments: dietary, activity, sleep assessment questionnaire, stress-related eating, 7-10-day accelerometer (activity, sleep), 7-10-day continuous glucose monitor

Genetic/ Epigenetic

* Genome-wide genotyping array
* Genome-wide DNA methylation array

Five-point MACE

* Acute myocardial infarction
* Stroke
* Cardiovascular mortality
* Hospitalization for unstable angina or revascularization procedures
* Heart failure

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet the following criteria according to their group:

Four categories of participants will be included in this study and the inclusion criteria for each group are given below:

* Participants with Y-T2DM

  * Age 12-25 years
  * Type 2 diabetes mellitus as defined by fasting blood glucose >= 126 mg/dL OR postprandial blood sugar >= 200 mg/dL OR Hemoglobin A1c >= 6.5 percent per American Diabetes Association Criteria OR documentation of type 2 diabetes diagnosed at <=25 years of age
* Youth with overweight/ obesity (Y-OW)

  * Age 12-25 years
  * For participants < 18 years of age, BMI >= 85th percentile (overweight) and >= 95th percentile (obesity) for age and sex OR
  * For participants >= 18 years of age, BMI >=25<30 kg/m^2 (overweight) or >=30 kg/m^2 (obesity)
  * Participants with obesity may have a diagnosis of prediabetes, defined as fasting blood glucose 100-125 mg/dL OR postprandial blood sugar 140-199 mg/dL OR HbA1c 5.7-6.4 percent (either during testing at NIH or as previously documented on outside medical record).
* Healthy control lean participants (Y-Lean)

  * Age 12-25 years
  * For participants < 18 years of age, BMI <= 85th percentile for age and sex OR
  * For participants >=18 years of age, BMI 18-24.99 kg/m^2.
  * HbA1c <5.7 percent (either during testing at NIH or as previously documented on outside medical record).
* Biological parents of Y-T2DM, Y-OW and Y-Lean participants

  * Biological parent of enrolled Y-T2DM, Y-OW and Y-Lean by self-report.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria for their specific group will be excluded from participation in this study:

* Y-T2DM, Y-OW and Y-Lean Participants:

  * Type 1 diabetes or the presence of >2 diabetes auto-antibodies (e.g., GAD-65, IA-2 antigen, Zinc transporter 8 autoantibodies).
  * Medical, psychiatric or cognitive disorders that will, in the opinion of the investigators, limit the subject s ability to comply with study procedures (specific obesity-related comorbidities are explicitly permitted, including hypertension, hyperlipidemia, obstructive sleep apnea and non-alcoholic steatohepatitis).
  * Serious medical illnesses or diseases thought to alter metabolism (including moderate to severe renal disease (< 30 mL/min/1.73m^2), congenital heart disease, Cushing s syndrome, cancer, or other metabolic diseases associated with diabetes or excess weight).
  * For participants enrolled at the NIH, dietary allergies, intolerances or eating patterns that would preclude them from consuming metabolic meals.
  * Unwilling to comply with all study procedures or to adhere to Lifestyle Considerations throughout study duration.
  * Pregnancy at the time of the screening visit.
  * Clinically significant anemia OR Hematocrit below the lower limit of normal for age and sex cutoffs.
* Y-Lean participants:

In addition to the above exclusion criteria, any Y-Lean participant who meets any of the following additional criteria will be excluded from the study:

* Current use of prescription or non-prescription medication. Certain exceptions are permitted, including topical medications, vitamins, and hormonal contraceptives. Other medications may be permitted at the discretion of the investigators.
* Recent (past 2 months) use of drugs or supplements that alter glucose or lipid metabolism (e.g., niacin, fish oil, red yeast rice)
* History of diabetes or abnormal glucose tolerance
* Abnormal screening labs, including the following:

  * ALT or AST >2 times the upper limit of normal
  * Glycosuria
  * Low eGFR (<90 mL/min/1.73m^2)Any other abnormality that, in the opinion of the investigator, will increase risk to the subject from participation, or interfere with interpretation of study data

    * Biological Parents
* No Exclusion Criteria

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will evaluate the pathophysiological features of cardiovascular disease in youth-onset type 2 diabetes (Y-T2DM) using a multi-level, multi-domain approach of socio-ecological risk factors (societal, community, and individual). We will employ a prospective, observational study design in youth aged 12-25 years to compare Y-T2DM with age and BMI-matched youth with overweight or obesity (Y-OW) and age-matched healthy lean peers (Y-Lean). The study will also include a single-day visit for biological parents of enrolled Y-T2DM, Y-OW and Y- lean, to assess parental factors involved in the pathophysiology of cardiovascular disease in Y-T2DM.
Sampling Method: Non-Probability Sample
Enrollment: 930 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2033-10-31 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity (PWV) | Baseline
  Carotid-femoral pulse wave velocity (m/s) measured with SphygmaCor, higher numbers indicated greater arterial stiffness
Augmentation index (Aix) | Baseline
  Augmentation index (%) measured with SphygmaCor, higher numbers indicated greater arterial stiffness.
Pulse wave velocity (PWV) | 5 Years
  Carotid-femoral pulse wave velocity (m/s) measured with SphygmaCor
Augmentation index (Aix) | 5 Years
  Augmentation index (%) measured with SphygmaCor

SECONDARY OUTCOMES:
Right coronary wall thickness | Baseline
  During cardiac MRI, cross-sectional analysis of right coronary artery vessel wall thickness; greater thickness associated with increased risk for endothelial dysfunction
Right coronary wall thickness | 5 years
  During cardiac MRI, cross-sectional analysis of right coronary artery vessel wall thickness; greater thickness associated with increased risk for endothelial dysfunction
Endothelial Function | Baseline
  During cardiac MRI, measurements of change in vessel wall thickness during isometric handgrip exercise. Smaller change associated with endothelial dysfunction
Endothelial Function | 5 years
  During cardiac MRI, measurements of change in vessel wall thickness during isometric handgrip exercise. Smaller change associated with endothelial dysfunction
Fasting remnant lipoproteins | Baseline
  Fasting plasma remnant lipoproteins measured with nuclear magnetic spectroscopy; higher concentrations associated with increased cardiovascular disease risk
Postprandial remnant lipoproteins | 5 years
  Plasma remnant lipoproteins measured with nuclear magnetic spectroscopy. Incremental area under the curve for plasma remnant lipoproteins will be calculated from the standard 5-hour mixed meal tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Chung, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - Children's National Hospital (CNH), Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide raw data (without identifying information) to journals or other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be provided upon request within 1 year after publication and will be available for at least 10 years
Access Criteria: The PI will accept requests from other researchers who are examining pertinent outcomes.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001819-DK.html